CLINICAL TRIAL: NCT00757679
Title: Evaluation of the Antinociceptive and Analgesic Effects of Milnacipran. An Exploratory Placebo-controlled Clinical Trial in Fibromyalgia Out-patients
Brief Title: Evaluation of the Antinociceptive and Analgesic Effects of Milnacipran
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F02207 GE 205
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Milnacipran (Experimental)
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — capsules
  Arms: Milnacipran
Drug: Placebo — capsules
  Arms: Placebo

SUMMARY:
Evaluation of the antinociceptive effect of 7 weeks of treatment with milnacipran, compared to placebo, in fibromyalgia out-patients

ELIGIBILITY:
Inclusion Criteria:

* patient with FMS according to the 1990 ACR criteria
* patient willing to withdraw from CNS-active therapies commonly used for FMS, including anti-depressants, anti-convulsivants, opiates
* patient willing to discontinue treatment with tender and trigger point injections, joint injections and anesthetics

Exclusion Criteria:

* severe psychiatric illness
* current Major Depressive Episode (MDE)
* significant risk of suicide
* history of substance abuse
* epilepsy
* myocardial infarction in the past 24 months
* active cardiac disease
* congestive heart failure
* prosthetic heart valve
* haemodynamically significant valvular heart disease
* known cardiac rhythm anomalies or conduction abnormalities
* unstable and uncontrolled arterial hypertension or supine arterial blood pressure over 160/90 mmHg
* pulmonary dysfunction
* active liver disease
* renal impairment
* documented autoimmune disease
* current systemic infection
* active cancer, except basal cell carcinoma or current cancer therapy
* severe sleep apnoea
* active peptic ulcer or inflammatory bowel disease (except IBS)
* unstable endocrine disease
* pregnancy or breastfeeding
* concomitant use of non selective MAO inhibitors, MAO-A or -B inhibitors, tricyclics, tetracyclics, SSRIs, NARIs, SNRIs, epinephrine, norepinephrine, clonidine and related compounds, long-acting benzodiazepines
* concomitant use of oral anticoagulants, anticonvulsants, type Ic antiarrythmics, lithium
* concomitant use of hypericum and SAMe
* concomitant use of digitalis preparations
* regular use of centrally-acting muscle relaxants
* concomitant use of strong analgesics, including tramadol, codeine or opiates
* any factor known to affect the HPA axis or autonomic function such as cigarette smoking (regularly over 25 cigarettes a day)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To assess the antinociceptive effect of 7 weeks of treatment with milnacipran, compared to placebo, in fibromyalgia outpatients. | 7 weeks

SECONDARY OUTCOMES:
The analgesic effect of 7 weeks of treatment with milnacipran, compared to placebo | 7 weeks
The correlation of the antinociceptive and analgesic effects of milnacipran with the cytochrome CYP2D6 and COMT phenotype polymorphism determinations | 7 weeks
The safety/tolerability and compliance of 8 weeks of treatment with milnacipran | 8 weeks
The therapeutic drug monitoring (TDM) and carry out the PK/PD correlations | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jules Desmeules, MD, Principal Investigator — Centre Hospitalier HUG Genève - SUISSE
Locations (1):
- Clinical Pharmacology & Toxicology Multidisciplinary Pain Centre, Geneva, Switzerland